CLINICAL TRIAL: NCT05552625
Title: Multicenter, Double-blind, Placebo-controlled, Maximum 10 Days Administration Study to Evaluate the Efficacy and Safety of TADIOS as an Adjuvant Therapy in Patients Diagnosed With Mild to Moderate COVID-19
Brief Title: The Efficacy and Safety of TADIOS as an Adjuvant Therapy in Patients Diagnosed With Mild to Moderate COVID-19
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This Phase I study was conducted in India and no subject data was provided to sponsor.
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 21PR0041-008
Record Dates: First submitted 2021-04-20; First posted 2022-09-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: COVID-19; Antioxidative biomarker; Inflammatory biomarker; TADIOS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TADIOS + Standard of care treatment (Active Comparator): 4 tablets of 300 mg each will be administered to the subjects twice daily (1200 mg in the morning and 1200mg in the evening making it 2400 mg/day) for a maximum of 10 days. The subject can consume standard of care treatment as per prescribed by the physician.
  Interventions: Drug: TADIOS
- Placebo + Standard of care treatment (Placebo Comparator): 4 tablets of 300 mg each will be administered to the subjects twice daily (1200 mg in the morning and 1200mg in the evening making it 2400 mg/day) for a maximum of 10 days. The subject can consume standard of care treatment as per prescribed by the physician.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TADIOS — TADIOS is a combination extract which composed of three herbs, and each herbal medicine has been traditionally used as a food or a herbal medicine treating various respiratory diseases in Asia
  Other Names: Herbs
  Arms: TADIOS + Standard of care treatment
Drug: Placebo — Combination of the following Lactose hydrate, Microcrystalline cellulose, Colloidal silicone dioxide, Povidone, Croscarmellose sodium, Magnesium stearate, Tabshield(79O245)
  Other Names: Lactose hydrate
  Arms: Placebo + Standard of care treatment

SUMMARY:
This study will assess the safety and efficacy and tolerability of TADIOS compared to placebo in patients with mild to moderate COVID-19.

DETAILED DESCRIPTION:
100 patients diagnosed with COVID-19 by RT-PCR were randomized in a ratio of 1:1 into TADIOS group and placebo group to evaluate efficacy and safety after intake over 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged between 18 to 65 years (both inclusive)
2. Confirmed Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) first infection by a reverse transcription polymerase chain reaction (RT-PCR) assay in nasal swab or oropharyngeal swab samples.
3. Patients who are hospitalized into designated hospital for COVID-19 treatment
4. Patients who can be treated within 24 hours after confirmed diagnosis with COVID-19
5. Patients with mild COVID-19 or moderate COVID-19 according to clinical management guideline of Government of India.

   * Mild Illness: Patients with uncomplicated upper respiratory tract viral infection, may have non-specific symptoms such as fever, cough, sore throat, nasal congestion, malaise, and headache. The elderly may present with atypical symptoms. These patients do not have any signs of dehydration, sepsis or shortness of breath.
   * Moderate Illness: Patient with pneumonia and no signs of severe pneumonia (Chest X-ray will be performed to rule out pneumonia in the suspected subjects).
6. Patients who have signed the written informed consent form approved by Ethics Committee to participate after understanding explanations regarding the study
7. Those who can comply with the requirements and processes in the clinical study
8. Women of childbearing age must be negative to urine pregnancy test during screening

Exclusion Criteria:

1. Patients with severe COVID-19
2. Self-reported history of meaningful circulatory, renal, gastrointestinal, liver, endocrinal, hematological, or mental disease, or other serious diseases or alcohol or drug addiction that may cause safety issues or confusion in the interpretation of clinical research results by the principal investigator's judgment
3. Female patients who are pregnant (confirmed through urine pregnancy test) or breastfeeding
4. Patients with cardiovascular, liver, cancer and kidney disease.
5. Self-reported patients being a recipient of immunosuppressive therapy
6. Self-reported patients who are allergic to this dietary supplements
7. Patients taking a health functional food or medicine that may affect the body's antioxidant, anti-inflammatory activity, and lungs within 6 weeks of the first visit
8. Patients who participated in another clinical trial within 1 month before screening
9. Patients have any condition that in the judgement of investigator make the subject inappropriate for entry into this study
10. Patients consuming any herbal medicine
11. Self-reported patients with cases of surgical menopause (hysterectomy, oophorectomy of both ovaries) or sterilization procedures (tubal ligation or tubectomy of both fallopian tubes). Menopause refers to 1 year of no menstruation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2022-02-24 (Estimated); Study Completion 2022-02-24 (Estimated)

PRIMARY OUTCOMES:
Evaluation of antioxidative and inflammatory Biomarkers | Day 1, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in Antioxidative and inflamatory biomarkers: TNF-α, CRP, IL-6, IL-1ra, Hb, and ferritin.
Clinical measurements - Ordinal Scale for COVID-19 Assessment | Day 1, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in Covid-19 8-point Ordinal Scale: 0 = Uninfected, 1 = Ambulatory without limitation of activity, 2 = Ambulatory with limitation of activity, 3 = Hospitalized mild disease, no oxygen, 4 = Hospitalized mild disease, supplemental oxygen, 5 = Hospitalized severe disease, non-invasive ventilation or high-flow oxygen, 6 = Hospitalized severe disease, intubation and mechanical ventilation, 7 = Hospitalized severe disease, ventilation plus additional organ support, 8 = Death.
Clinical measurements - Clinical Recovery Scale for COVID-19 Assessment | Every day from screening till discharge and Day 14 after last IP administration
  Time to clinical recovery in COVID-19 Clinical Symptom Scale: The clinical symptom scale has been designed for this study to access the clinical state and time taken to relieve the clinical symptoms of COVID-19 (fever, dry cough, tiredness, aches and pains, sore throat, diarrhea, headache, loss of taste, loss of smell, difficulty in breathing or shortness of breath and chest pain or pressure).
Clinical measurements Clinical Improvement Scale for COVID-19 Assessment | Daily from screening to discharge or Day 14 after last IP administration
  Proportion of Clinical Improvement in Clinical Symptom Scale (Count of subjects with and without a symptom by treatment group on each day with the previous day counts during the study period).
Assessment of Quality of life - WHO-5 Well-Being Index | Day 1, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in WHO-5 Well-Being Index: The total raw score, ranging from 0 to 25, will be multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Assessment of Quality of life - Fatigue Severity Score | Day 1, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in Fatigue Severity Score: Minimum total score possible is nine and the maximum is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities.
Hospitalization - Time to discharge | Day 1, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10)
  1. Duration of hospitalization
  2. Time to discharge

SECONDARY OUTCOMES:
Safety and tolerability assessment after administration of TADIOS 1 | Screening, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Subject incidence of Treatment-Emergent Adverse Events (TEAEs) and total number of unique TEAEs.
Safety and tolerability assessment after administration of TADIOS - Hematology | Screening, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in Hematology, Complete Blood Count results WBC, RBC, Hb, HCT, MCV, MCH, MCHC, PLT, MPV, differential count of WBC (Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil), and ESR.
Safety and tolerability assessment after administration of TADIOS - Serum Chemistry | Screening, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in Serum Chemistry results: total protein, albumin, globulin, A/G ratio, total bilirubin, AST, ALT, GGT, Random glucose, BUN, creatinine, estimated GFR, Ca2+, phosphate, Na+, K+, Cl-, CRP, triglyceride, cholesterol, HDL-cholesterol, and LDL-cholesterol.
Safety and tolerability assessment after administration of TADIOS - Urinalysis | Screening, Maximum Day 10 (The date of discharge or early termination, from Day 1 to Day 10) and Day 14 after last IP administration
  Change from baseline in Urinalysis results: Color, pH, Specific gravity, albumin, bilirubin, glucose, urobilinogen, ketone, nitrite, hematuria, leukocyte and microscopy.
Safety and tolerability assessment after administration of TADIOS - Blood Pressure | Screening, Maximum Day 10 (The date of discharge or early termination, at Day 1, 2, 4, 7, 10) and Day 14 after last IP administration
  Change from baseline in Blood Pressure in mm Hg.
Safety and tolerability assessment after administration of TADIOS - Body Temperature | Screening, Maximum Day 10 (The date of discharge or early termination, at Day 1, 2, 4, 7, 10) and Day 14 after last IP administration
  Change from baseline in Body Temperature ℃.
Safety and tolerability assessment after administration of TADIOS - Pulse Rate | Screening, Maximum Day 10 (The date of discharge or early termination, at Day 1, 2, 4, 7, 10) and Day 14 after last IP administration
  Change from baseline in Pulse Rate in beats per minute.
Safety and tolerability assessment after administration of TADIOS - Respiration Rate | Screening, Maximum Day 10 (The date of discharge or early termination, at Day 1, 2, 4, 7, 10) and Day 14 after last IP administration
  Change from baseline in Respiration Rate in breaths per minute.

CONTACTS AND LOCATIONS:
Overall Officials: John M Paul, MD, Principal Investigator — Sparsh Hospital
Locations (6):
- India (6):
  - Vagus Super Specialty Hospital, Bangalore, Karnataka
  - Sparsh Superspeciality Hospital, Bangalore, Karnataka
  - Lakshmi Nursing Home, Kochi, Kerala
  - Chaitanya Hospital, Paravūr, Kerala
  - Gunjkar Multispeciality Hospital, Pune, Maharashtra
  - Oxycare Multispecialty Hospital, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No